CLINICAL TRIAL: NCT00690092
Title: Safety, Sensitivity and Specificity of Spherule-derived Coccidioidin in Naive Adults, in Adults With a History of Pulmonary Coccidioidomycosis and in Adults With a History of Pulmonary Histoplasmosis
Brief Title: A Multi-center Study of Spherule-Derived Coccidioidin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nielsen BioSciences, Inc. (Industry)
Collaborators: Sr Consultants Inc. (Industry)
Responsible Party: Harry S. Nielsen, Ph.D., Allermed Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: S104-1, S104-2, S104-3
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Coccidioidomycosis
Keywords: Coccidioidin; Coccidioidin SD; Spherule-derived coccidioidin; Coccidioidomycosis; Valley Fever; Coccidioides immitis
MeSH Terms: conditions — Coccidioidomycosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Volunteers with a history of pulmonary coccidioidomycosis verified by serology and/or histology or mycology.
  Interventions: Biological: Spherule-derived coccidioidin
- 2 (Active Comparator): Volunteers without a history of pulmonary coccidioidomycosis confirmed by serology (naive).
  Interventions: Biological: Spherule-derived coccidioidin
- 3 (Active Comparator): Volunteers with a history of pulmonary histoplasmosis but no history of coccidioidomycosis confirmed by serology.
  Interventions: Biological: Spherule-derived coccidioidin

INTERVENTIONS:
Biological: Spherule-derived coccidioidin — 1.27 ug of sterile, injectable product (spherule-derived coccidioidin). Product was administered once by intradermal injection along with positive and negative control agents and results read after 48 hours.
  Other Names: Coccidioidin SD (proposed trade name)

SUMMARY:
Adult volunteers were skin tested with 1.27 ug spherule-derived coccidioidin. The skin test antigen was evaluated in three different populations of adult volunteers to determine the safety and efficacy of the product in the assessment of delayed-type hypersensitivity to Coccidioides immitis. Induration greater than or equal to 5 mm after 48 hours was considered positive for exposure to C. immitis.

ELIGIBILITY:
Inclusion Criteria:

* Good Health (absence of active medical disease)
* Meets criteria specific to population groups:

  * Coccidioidomycosis Group:
* History of coccidioidomycosis of at least 45 days duration confirmed by roentgenograph serologic or mycologic findings

  * Histoplasmosis Group:
* History of pulmonary histoplasmosis

  * Naive Control Group:
* Lifetime residence in the states of WA, OR, ID, or MT
* Never employed as an agricultural worker
* Serology negative for C.immitis antibodies

Exclusion Criteria (All Groups):

* Active medical disease
* Alcohol abuse or illicit drug use
* Influenza-like illness within the past 4 weeks
* Immunizations within the past 4 weeks
* Current atopic or contact dermatitis, psoriasis, erythema nodosum, urticaria
* Current treatment with corticosteroids, cytotoxic or immunosuppressive drugs
* Immunodeficiency disease
* HIV infection
* Previous skin test with coccidioidin or SD Coccidioidin
* Pregnant or lactating
* Adverse reaction to thimerosal
* Adverse reaction to Candida or Trichophyton skin test antigens

Coccidioidomycosis Group:

* Current cavitary or disseminated coccidioidomycosis
* History of histoplasmosis, or blastomycosis

Histoplasmosis Group:

* History of coccidioidomycosis or blastomycosis

Naive Control Group:

* History of coccidioidomycosis, histoplasmosis, blastomycosis
* Travel for more than 30 days in designated areas of CA, AZ, NV, UT, NM, TX and Mexico, Central and South America. Travel for more than 7 days in restricted areas of CA, AZ and TX.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2005-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To determine the ability of spherule-derived coccidioidin to detect cellular hypersensitivity to C. immitis by a positive DTH skin test in a population with a history of pulmonary coccidioidomycosis. | 48 hours

SECONDARY OUTCOMES:
Determine the specificity of spherule-derived coccidioidin by testing the skin test antigen in naive adult volunteer and volunteers with a history of pulmonary histoplasmosis. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Harry S Nielsen, Ph.D., Study Director — Nielsen BioSciences, Inc.; Royce Johnson, M.D., Principal Investigator — Kern Medical Center; Neil Ampel, M.D., Principal Investigator — University of Arizona, Tucson; Brad Sawtelle, M.D., Principal Investigator — Blair, NE; Stephen Kernerman, D.O., Principal Investigator — Spokane, WA
Locations (4):
- United States (4):
  - Health Sciences Center AVAHCS, Univ. of Arizona, Tucson, Arizona
  - Kern Facility Medical Group, Bakersfield, California
  - Blair Clinic, Blair, Nebraska
  - Spokane Allergy and Asthma Center, Spokane, Washington